CLINICAL TRIAL: NCT02888639
Title: EPHEYL: Étude PHarmacoÉpidémiologique de l'hYperparathyroïdie Secondaire en Lorraine
Brief Title: Pharmacoepidemiological Study of Secondary Hyperparathyroidism in Lorraine
Acronym: EPHEYL
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: EPHEYL
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The pharmacoepidemiological EPHEYL (Étude PHarmacoÉpidémiologique de l'hYperparathyroïdie secondaire en Lorraine) study is a 2-year, open-cohort, prospective, observational study on incident SHPT, i.e. newly diagnosed, with a 2 year follow-up, set in the 12 dialysis units located in the French region of Lorraine (public or private).

DETAILED DESCRIPTION:
In the early stages of the disease, 90% of patients with chronic renal failure present evidence of bone remodeling due to secondary hyperparathyroidism (HPT). As the disease progresses and patients require dialysis for end-stage renal failure (ESRF), the incidence of secondary HPT declines to 25-40% with reduced bone remodeling as shown by osteomalacia observed in 4-12% of patients and adynamic bone in 20-40%. Observational studies have described an association between serum phosphorus level, phosphorus-calcium product, parathormone (PTH) level, and mortality. Since there is no real consensus, treatments, basically diet and drugs, are tailored to each individual. The therapeutic range is wide and interactions are frequent. Therapeutic efficacy is compromised by the variability of PTH assay results, the ambulatory nature of interventions, and poor patient adherence. The guidelines issued in 2003 stipulate that corrective measures, i.e. dietetic counseling with or without drug therapy, are needed when serum PTH exceeds 300 pg/ml. When the PTH level exceeds 500, or even more so 800 pg/ml, HPT can constitute an indication for parathyroid surgery or calcimimetic treatment.

Data from a randomized comparison between cinacalcet and surgery are lacking. The evidence-based decision for surgery is made conjointly by the nephrologist, the surgeon and the patient, limiting the feasibility of randomization. Parathyroidectomy can be achieved by three techniques whose efficacy has been studied in historical observational studies. Cinacalcet received marketing approval in 2004 for "the treatment of secondary HPT in patients with ESRF treated by dialysis. Mimpara can be used in the context of a regimen including phosphate chelators and/or vitamin D analogs, as needed". Four double-blind studies have demonstrated the efficacy of cinacalcet versus placebo in decreasing the PTH level, but there is no proof of the efficacy of cinacalcet in terms of cardiovascular events and mortality. One cost-effectiveness study showed that parathyroidectomy was superior to cinacalcet, except if the patient was on dialysis for a short period before renal transplantation or presented contraindications for surgery.

While randomized trials are the gold standard, such trials include a limited number of patients for a limited period of time. This does not enable an observation of long-term practices and adverse effects. Moreover, such trials do not concern patients with other co-morbid conditions taking several drugs, in particular, elderly subjects. The concept of the pharmacoepidemiological study is to describe real-life populations taking a given drug, using both quantitative and qualitative parameters to determine efficacy, risk, and drug use in real-life conditions free of the constraints of a clinical trial.

ÉPHÉYL is an observational pharmacoepidemiological study concerning the prescription of calcimimetic agents and parathyroidectomy in patients with ESRF on dialysis who present severe secondary HPT (PTH ≥ 500 pg/ml). The aim is to describe indications and efficacy: control of PTH, calcium and phosphorus serum levels within their recommended ranges, patient tolerance of the therapeutic interventions, and the cost of such interventions, as well as patients' adhesion to treatment and their self-assessed quality-of-life. This three-year inclusion study, based on the Lorraine REIN registry, will involve all participants in the Néphrolor network. The study will begin on April 1st, 2009.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* Patient on hemodialysis or peritoneal dialysis for 3 months or more in one of the 12 dialysis units in the study.
* Patient included in the REIN registry in the Lorraine region.
* Parathormone greater than or equal to 500 pg / ml for the first time after 01/04/2009 (patient incident for secondary hyperparathyroidism).

Exclusion Criteria:

* age < 18 years.
* Patient living in Lorraine but dialysed in a unit outside Lorraine.
* Diagnosis of secondary hyperparathyroidism with higher parathormone or equal to 500 pg / ml placed before 1/4/2009.
* Patient who have received medical treatment with cinacalcet or by surgical parathyroidectomy for secondary hyperparathyroidism.
* Patient expressing opposition to the collection of information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD requiring mainteance dialysis
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Parathormone level | 2 years
  Obtaining the therapeutic target according to the K/DOQI

SECONDARY OUTCOMES:
Phosphocalcium product level | 2 years
Serum calcium level | 2 years
Serum phosphorus level | 2 years
Symptoms and / or clinical events caused by hyperparathyroidism | 2 years
  using clinical and paraclinical examinations
Tolerance of therapeutic interventions: nausea, vomiting, diarrhea, hypocalcemia | 2 years
  using clinical and paraclinical examinations
The quality of life | 2 years
  using the KDQOL questionnaire
Satisfaction of professionals | 2 years
  Interview of professionals on patient care
The direct costs of treatment | 2 years
  Cost related to medical treatment, parathyroidectomy, hospitalisation, clinical and paraclinical examination
Patient compliance | 2 years
  using the CET (Compliance Evaluation Test ) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luc Frimat, MD, PhD, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filipozzi P, Ayav C, Ngueyon Sime W, Laurain E, Kessler M, Brunaud L, Frimat L. Trajectories of CKD-MBD biochemical parameters over a 2-year period following diagnosis of secondary hyperparathyroidism: a pharmacoepidemiological study. BMJ Open. 2017 Mar 27;7(3):e011482. doi: 10.1136/bmjopen-2016-011482. PMID 28348181